CLINICAL TRIAL: NCT04176653
Title: Phase 1b Single Ascending and Multiple Dose First-in-man Study in Adult Patients With Non-transfusion-dependent Beta-thalassaemia or Low Risk Myelodysplastic Syndrome to Investigate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Response of SLN124
Brief Title: Study in Beta-thalassaemia or Myelodysplastic Syndrome Patients to Investigate the Safety and Tolerability of SLN124
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopped prior to subject administered first dose, due to COVID-19
Sponsor: Silence Therapeutics plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLN124-001
Record Dates: First submitted 2019-11-07; First posted 2019-11-25 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Non-transfusion-dependent Thalassemia; Low Risk Myelodysplastic Syndrome

STUDY DESIGN:
Intervention Model Description: Multiple Group Assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: SLN124 is a GalNAc conjugated double stranded fully modified siRNA. Sodium chloride 0.9% w/v is used as Placebo
- 0.3 mg/kg (Experimental)
  Interventions: Drug: SLN124 is a GalNAc conjugated double stranded fully modified siRNA. Sodium chloride 0.9% w/v is used as Placebo
- 1.0 mg/kg (Experimental)
  Interventions: Drug: SLN124 is a GalNAc conjugated double stranded fully modified siRNA. Sodium chloride 0.9% w/v is used as Placebo
- 3.0 mg/kg (Experimental)
  Interventions: Drug: SLN124 is a GalNAc conjugated double stranded fully modified siRNA. Sodium chloride 0.9% w/v is used as Placebo
- 10.0 mg/kg (Experimental)
  Interventions: Drug: SLN124 is a GalNAc conjugated double stranded fully modified siRNA. Sodium chloride 0.9% w/v is used as Placebo

INTERVENTIONS:
Drug: SLN124 is a GalNAc conjugated double stranded fully modified siRNA. Sodium chloride 0.9% w/v is used as Placebo — IMP will be provided as a solution to be injected by qualified clinical staff in patient's abdomen, upper arms or front of the thighs.

SUMMARY:
The primary purpose of this study is to determine the safety and tolerability of SLN124 for the treatment of non-transfusion-dependent (NTD) β-thalassaemia and low risk myelodysplastic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18yrs; BMI 18-35 kg/m2
* β-thalassaemia intermedia or compound heterozygous HbE/β-thalassaemia
* Non-transfusion dependent: ≤ 5 units red cells in last 6 months and transfusion-free for ≥8 weeks
* Hb between 5 & 11 g/dL
* Ferritin > 250 µg/L and /or liver iron ≥ 3mg Fe/g dry weight and TSAT >40%

Exclusion Criteria:

* Haemoglobin S/β-thalassaemia, homozygous β-0 thalassaemia or α thalassaemia
* ALT/AST > 1.5 x upper limit normal or cirrhosis
* eGFR < 60 mL/min/1.73m2
* Platelets <100 or > 1000 x 109/L
* Untreated B12/folate deficiency
* Iron chelation therapy unless stable for ≥8 weeks
* Daily NSAID, therapeutic dose anticoagulant, ESA ≤12 weeks or stable dosing of hydroxyurea ≤ 6 months
* Significant cardiac disease (MI in 6 months, NYHA class III-IV heart failure, long QT)
* HIV or active hepatitis B/C or malignancy within 5 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-10-14 (Estimated)

PRIMARY OUTCOMES:
# of participants with all AEs as assessed by CTCAE V4.0 included injection site reaction, will be measured from baseline to post dose follow up | Up to two months
12 lead electrocardiogram parameters included PR, QTcF and QTcB will be measured from baseline to post dose follow up | Up to two months
clinical chemistry, haematology, urinalysis, liver function tests (included ALT, AST, GGT) will be measured from baseline to post dose follow up | Up to two months
height, weight, blood pressure, heart rate, respiration rate and temperature will be measured from baseline to post dose follow up | Up to two months

SECONDARY OUTCOMES:
Biomarkers will be measured from baseline to post dose follow up | Up to two months
  serum hepcidin level (ng/ml), ferritin level (ug/L), Transferrin saturation (%), iron level (umol/L), haemoglobin and reticulocyte count will be analysed by central laboratory.
Pharmacokinetic of SLN124 in plasma from baseline to post dose follow up | Up to two months
  Peak Plasma Concentration (Cmax) will be analysed by central laboratory.
Pharmacokinetic of SLN124 in plasma from baseline to post dose follow up | Up to two months
  Area under the plasma concentration versus time curve (AUC) will be analysed by central laboratory.

CONTACTS AND LOCATIONS:
Locations (5):
- Bulgaria (4):
  - MHAT Dr. Nikola Vasiliev AD, Kyustendil
  - UMHAT Dr. Georgi Stranski AD, Pleven
  - Medical Center COMAC MEDICAL, Sofia
  - UMHAT Sv. Ivan Rilski, Sofia
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No